CLINICAL TRIAL: NCT05894980
Title: Controlled Randomized Non-comparative Trial Assessing Active Transcranial Direct Current Stimulation [tDCS] on Left Dorsoleteral Prefrontal Cortex Versus Active tDCS Active on Right Orbitofrontal Cortex to Treat Unipolar Depression
Brief Title: How to Reduce Suicidal Thoughts and Impulsivity in Depression
Acronym: DEPIMPULSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Fondation FondaMental (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/724
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Unipolar Depression; Impulsive Behavior; Suicidal Ideation
Keywords: transcranial stimulation; tDCS; left PreFrontalDorsoLateral Cortex; right OrbitoFrontal Cortex
MeSH Terms: conditions — Depressive Disorder; Impulsive Behavior; Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active tDCS on left DLPFC (Experimental): Active tDCS applied on left dorsolateral prefrontal cortex [DLPFC]
  Interventions: Device: active tDCS stimulating left DLPFC
- active tDCS on right OFC (Active Comparator): Active tDCS applied on right orbitofrontal cortex [OFC]
  Interventions: Device: active tDCS stimulating right OFC
- sham tDCS (Sham Comparator): Sham tDCS applied on left dorsolateral prefrontal cortex [DLPFC]
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS stimulating left DLPFC — 20 active tDCS sessions (4 sessions/day for 5 days, 30 min each, 2 mA) applied to the left DLPFC
  Other Names: Starstim® (Neuroelectrics, Spain)
  Arms: active tDCS on left DLPFC
Device: active tDCS stimulating right OFC — 20 active tDCS sessions (4 sessions/day for 5 days, 30 min each, 2 mA) applied to the right OFC
  Other Names: Starstim® (Neuroelectrics, Spain)
  Arms: active tDCS on right OFC
Device: sham tDCS — 20 active tDCS sessions (4 sessions/day for 5 days, 30 min each, 0 mA) applied to the left DLPFC
  Other Names: Starstim® (Neuroelectrics, Spain)
  Arms: sham tDCS

SUMMARY:
The study aims at investigating if tDCS applied to left DLPFC or to right OFC to treatment as usual is effective in reducing severe suicidal ideas in major depressive episode.

DETAILED DESCRIPTION:
Depressive disorders are one of the most frequent pathologies in psychiatry. The lifetime prevalence of the characterized depressive episode is indeed particularly high, between 16.6% in the United States and 24.1% in France. Because of this high prevalence, and because they constitute a pathology with a high risk of suicidal behavior (SC), depressive disorders are a major target of medical strategies for suicide prevention. In addition to suicidal ideation, impulsivity, considered as the tendency to express spontaneous, excessive and/or unplanned behaviors, is recognized as being a major factor precipitating SCs.

With a pilot, prospective, multicenter design, the perspectives of DEPIMPULSE include being able to develop an innovative therapeutic approach in the reduction of risky behaviors, in particular suicidal ideation, associated impulsivity, suicidal risk in patients suffering from depression, while improving our understanding of the behavioral aspects and associated cognitions.

The treatment will be delivered during 5 consecutive days (D1 to D5).

Baseline measures (D0) will be compared to those obtained after the treatment administration (last day of treatment (D5) and 2 weeks (+W2) and 1 month (+W4) after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman older than 18 years oldRight-handed
* Signed Informed Consent form
* Subject affiliated to or beneficiary from a French social security regime
* Inpatient or outpatient at the Adult Psychiatry Service
* Diagnosis of Major Depressive Disorder according to the 5th edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria and confirmation by the MINI Structured Clinical Interview
* MADRS score ≥ 18
* Beck Scale for Suicide Ideation (BSS) score ≥8
* Under antidepressant treatment
* Absence of severe progressive neurologic and/or somatic pathologies (specially tumors, degenerative diseases)

Exclusion Criteria:

* tDCS contraindication
* Younger than 18 years old
* Left-handed
* under mood stabilizer and/or antiepileptic
* treated by ECT or rTMS or tDCS for the current eposide
* Subject under measure of protection or guardianship of justice
* Presence of other psychiatric pahtologies
* Subject beneficiary from a legal protection regime
* Subject unlikely to cooperate or low cooperation stated by investigator
* Subject not covered by social security
* Pregnant woman
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
BSS scores | Baseline (Day 0), Day 5 (D5)
  Difference of Beck's Scale for Suicide Ideation [BSS] score between Day 0 and Day 5, and between the arm active tDCS on left DLPFC and the arm active tDCS on right COF.
  This scale contains 19 items to assess the risk level for suicide among general population. French version of this scale is designed for autovaluation.
  Each item is quoted from 0 (no suicidal thoughts) to 2 (high degrees of suicidal intent).

SECONDARY OUTCOMES:
BSS scores | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Difference of Beck's Scale for Suicide Ideation [BSS] score between Day 0 and Day 5, +W2 and +W4 between the 3 arms This scale contains 19 items to assess the risk level for suicide among general population. French version of this scale is designed for autovaluation.
  Each item is quoted from 0 (no suicidal thoughts) to 2 (high degrees of suicidal intent).
C-SSRS scores | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Compared scores from the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS is a clinician-rated tool that evaluates suicidal ideation and behavior. It is composed by 6 "yes/no" questions. High suicide risk is indicated when "yes" is answered to questions 4, 5 or 6.
BIS-10 scores | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Compared scores from the French version of the Barratt Impulsiveness Scale (BIS-10). The French version of the BIS-10 is a self-rated 34 item questionnaire, composed by three subscales: motor-impulsivity, cognitive-impulsivity and non-planning-impulsivity. Each item is scored on a 0 to 4 points scale. Higher scores indicate higher levels of impulsivity.
UPPS scores | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Compared scores from the Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency Impulsive Behavior Scale (UPPS-P). The French version of the UPPS-P is a self-rated 45 item scale, evaluating the following components: urgency, lack of premeditation, lack of perseverance and sensation seeking. Each item is scored on a base of 4 points. Higher scores indicate higher levels of impulsivity.
BART scores | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Balloon Analogue Risk Task (BART), assessing risk-taking behavior
Cognitive assessment | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Compared results from the experimental TEA, assessing cognitive functions.
Delay discounting with MCQ scores | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Compared scores from the French version of the Monetary Choice Questionnaire (MCQ). The MCQ is a self-rated 27 item questionnaire which assessed the discounting. Delay discounting is the decline in the present value of a reward with delay to its receipt.
  Example item: " Would you prefer 25€ today or 75€ in 15 days? " For each item, subjects must choose between a low immediate reward and a higher delayed reward.
  Waiting times vary from 7 days to 186 days, and rewards are divided into 3 magnitudes: low (25-35€), medium (50-60€), high (75-85€).
  This will allow assessing: the influence of the the magnitude of the difference between the two rewards proposed, the impact of the time on the reward's subjective value (speed at which the reward is devalued over time), reflected in the k index.
  This index is calculated separately for each magnitude, and an average index is calculated for each subject.
  The more the k index is high, the more the subject is considered impulsive.
Severity of depressive symptoms evaluated by the clinician | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Score achieved on the validated clinician questionnaire Quick Inventory of Depressive Symptomatology (QIDS-C16) evaluating the severity of depressive symptoms.
  The QIDS-C16 was derived from specified items in the IDS-C30, clinician-rated scale to assess the severity of a participant's depressive symptoms. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
Severity of depressive symptoms evaluated by the patient | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Score achieved on the validated self-reported (QIDS-SR16) evaluating the severity of depressive symptoms. QIDS-SR-16 is a standard questionnaire "The Quick Inventory of Depressive Symptomatology" (16-Item) (Self-Report). This covers questions on falling asleep, sleep during the night, waking up , sleeping too much, feeling sad ,appetite, weight, concentration , how they view themselves, thoughts of death and suicide, general interests, energy levels, feeling slowed down , feeling restless.
Quality of life measured with the EQ-5D-5L | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Quality of life measured with the EQ-5D-5L
Psychological and Physical Pain-Visual Analogic Scale (PPP-VAS) | Baseline (Day 0), Day 5 (D5), Week 2(+W2) and Week 4 (+W4) post-tDCS
  Likert scales from 0 (none) to 10 (maximum possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Djamila BENNABI, MD PhD, Principal Investigator — CHU de Besançon
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Chenevier, GH Henri Mondor, Créteil
  - CHU de Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No